CLINICAL TRIAL: NCT03119116
Title: Pattern of Use of Direct Oral Anticoagulants in Non-valvular Atrial Fibrillation Patients in UK General Practices
Brief Title: Use of Direct Oral Anticoagulants in UK
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19330
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Stroke
Keywords: Stroke Prevention in NVAF patients
MeSH Terms: conditions — Stroke | interventions — Rivaroxaban; Dabigatran; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stroke Prevention with Rivaroxaban in NVAF Patients: All NVAF patients above 18 years for age prescribed with Rivaroxaban during the study period
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Stroke Prevention with Dabigatran in NVAF Patients: All NVAF patients above 18 years for age prescribed with Dabigatran during the study period
  Interventions: Drug: Dabigatran
- Stroke Prevention with Apixaban in NVAF Patients: All NVAF patients above 18 years for age prescribed with Apixaban during the study period
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Oral direct factor Xa inhibitors, 15mg and 20mg tablets QD
  Groups: Stroke Prevention with Rivaroxaban in NVAF Patients
Drug: Dabigatran — Oral direct thrombin inhibitors, 75mg and 150mg capsules BID
  Groups: Stroke Prevention with Dabigatran in NVAF Patients
Drug: Apixaban — Oral direct factor Xa inhibitors, 2.5mg and 5 mg tablets BID
  Groups: Stroke Prevention with Apixaban in NVAF Patients

SUMMARY:
Many people who suffer from irregular heartbeats (atrial fibrillation) which might cause stroke, need to take blood thinners to prevent it. It is important to prescribe the correct dose of blood thinners to the right patients to ensure the treatment works however avoiding complications. In the recent years, new blood thinners have been available; they require less laboratory tests and fewer visits to a doctor compared to older therapies. This study will look at how the general practitioners in the UK prescribe blood thinners according to the instructions given by the product manufacturer. We will use primary care data that is routinely collected by the general practitioners about their patients but without any possibility to identify individual patients. The results will help us to understand the magnitude of deviation from instructions in order to ensure that the patients benefit from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >= 18 years with at least one year of enrollment with the primary care practice and one year since first health contact recorded in the database THIN(The Health Improvement Network) or CPRD(Clinical Practice Research Datalink) prior to index prescription date will be included.
* Patients with first prescription of DOACs (rivaroxaban, dabigatran, apixaban) during the study period.
* Diagnosis NVAF (any time prior index date or within the 2 weeks after the index date)

Exclusion Criteria:

* Patients having the history of valvular replacement or mitral stenosis (prior to index date or 2 weeks after index-date)
* Patients who have any record of being prescribed their index drug prior to the enrolment period or who qualify as members of more than one cohort on the same day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based on primary care databases representative of the UK population.
Sampling Method: Non-Probability Sample
Enrollment: 31336 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Demographic Characteristics | 6 years
  * Age
  * Sex
  * Smoking status (previous 6 months)
  * Body mass index (previous 6 months)
  * Blood pressure history (previous 12 months)
  * Number of patients that are naïve vs non-naïve For non-naïve: type and duration of anticoagulant used before index date
Risk factor categories | 6 years
  * C(Congestive heart failure) H(Hypertension)A(Age)D(Diabetes Mellitus)S2(Prior Stroke or TIA) score
  * C(Congestive heart failure) H(Hypertension)A2(Age ≥75 years)D(Diabetes Mellitus)S2 V(Vascular disease)A(Age 65-74 years)SC(Sex category)
  * H(Hypertension)A(Abnormal renal and liver function)S(Stroke)B(Bleeding)L(Labile INRs)E(Elderly)D(Drugs or alcohol) score
  * INR(International Normalized Ratio) measurement
Previous medical history | 12 months prior to index date
  * Acute MI(Myocardial Infarction)
  * Stroke or TIA(Transient Ischemic Attack)
  * Systemic peripheral arterial embolism
  * Coronary artery disease
  * Congestive heart disease
  * Hypertension
  * Diabetes Renal disease (eGFR) or ACR (Albumin/Creatinine Ratio)
Previous medication history | 12 months prior to index date
  * Anti-arrhythmics
  * Statins
  * Anti-platelets
  * Beta-blockers
  * ACE(Angiotensin-Converting-Enzyme) inhibitors
  * Anti-diabetic agents
  * Non-steroidal anti-inflammatory drugs (NSAIDs)
  * Antacids
  * Histamine receptor antagonists
  * Proton pump inhibitors (PPIs)
  * Disease-modifying anti-rheumatic drugs (DMARDs)
  * Antidepressants
  * Antipsychotic agents
  * Oral contraceptives
  * Hormone replacement therapy (HRT)
  * Strong inhibitors of Cytochrome P450 or P-GP
  * Strong inducers of CYP3A4
Previous use of VKA | Ever prior to index date
  * Warfarin
  * Other Vitamin K antagonist(s)
Concurrent co-medication | 6 years
  * Anti-coagulants
  * Aspirin
  * Clopidogrel
  * Other
Daily dose | 6 years
  DOACs(new oral anticoagulants ) for stroke prevention in NVAF(Non valvular Atrial Fibrillation) patients including those with renal impairment
Dose posology | 6 years
  DOACs for stroke prevention in NVAF patients including those with renal impairment
Naive status and Non-naive status | 6 years
  DOACs for stroke prevention in NVAF patients including those with renal impairment
Treatment Duration | 6 years
  DOACs for stroke prevention in NVAF patients including those with renal impairment

SECONDARY OUTCOMES:
Time-trends | 6 years
  Characteristics of first-time use of DOACs in NVAF patients

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/